CLINICAL TRIAL: NCT07249190
Title: A Study to Evaluate the Safety and Effectiveness of Magnetic Resonance-Guided Ultrasound Ablation of the Anterior Nucleus of Thalamus for the Treatment of Drug-resistant Epilepsy.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Longsheng Pan, PLA General Hospital, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 301EP
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Epilepsy (Treatment Refractory)
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: MRgFUS treating epilepsy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MR-guided Focused Ultrasound Treating Epilepsy (Experimental)
  Interventions: Procedure: MR-guided Focused Ultrasound Therapy

INTERVENTIONS:
Procedure: MR-guided Focused Ultrasound Therapy — MR-guided Focused Ultrasound Therapy focusing Anterior Nucleus of the thalamus

SUMMARY:
The study "Safety and Efficacy Evaluation of MR-Guided Focused Ultrasound Anterior Thalamic Nucleus Ablation for Drug-Resistant Epilepsy" from Chinese PLA General Hospital, is a single-center, prospective, single-arm study. It uses a MR-guided Focused Ultrasound Therapy System and plans to recruit 20 patients with drug-resistant epilepsy who are ≥20 years old, have a WAIS score ≥70, an average of ≥3 monthly epileptic seizures in the 3 months before enrollment, and are refractory to at least 2 antiepileptic drugs (including 1 first-line drug), excluding those with unstable cardiac function, brain tumors, previous brain surgery history, etc. Anterior thalamic nucleus ablation is performed via MRgFUS, with multiple follow-ups from 48 hours to 2 years postoperatively. Safety is evaluated by the incidence of adverse events within 2 years, efficacy by seizure frequency recorded in epilepsy diaries and the QOLIE-31 scale. Statistical analysis is conducted using toolkits, while risks such as MRI-induced claustrophobia and CT radiation are controlled. It adheres to GCP and the Declaration of Helsinki to ensure data authenticity and subjects' rights. The technology provider is responsible for the normal operation of the device and providing 20 sets of treatment consumables.

ELIGIBILITY:
Inclusion Criteria:

Male or female aged no less than 20 years old; Capable of signing the informed consent form and able to attend all study visits; Diagnosed as drug-resistant epilepsy by an epilepsy specialist; The subject's epilepsy is ineffective to the adequate use of at least two antiepileptic drugs, one of which must be a first-line drug. Adequate drug use is defined as the therapeutic dose of each drug or the occurrence of side effects with the increase of drug dose; Capable of communicating during the operation; Wechsler Adult Intelligence Scale (WAIS) score ≥ 70; The average number of epileptic seizures is ≥ 3 per month within 3 months before enrollment. The drug dose remains stable within 3 months before enrollment; The anterior nucleus of thalamus is identifiable on MRI (structural T1 and T2 images); Willing and able to keep an epileptic seizure diary.

Exclusion Criteria:

The frequency of epileptic seizures is < 3 times per month within 3 months before the subject is enrolled; The subject's Wechsler Adult Intelligence Scale (WAIS) score < 70; The subject cannot maintain the drug dose within 3 months after receiving treatment; The subject has epilepsy caused by previous infection (such as herpes virus); The subject has idiopathic epilepsy (Lennox-Gastaut syndrome, drop attacks); The subject is pregnant or lactating;

The subject has the following manifestations of unstable cardiac function:

1. Unstable angina pectoris under medication;
2. Medical records of myocardial infarction within 6 months before entering the study;
3. Congestive heart failure that is not effectively controlled or is deteriorating;
4. History of arrhythmia with hemodynamic disturbance;
5. Patients with implanted cardiac pacemakers;
6. Severe hypertension (diastolic blood pressure still > 100 mmHg after drug control); The subject exhibits behaviors consistent with alcohol addiction or substance abuse; History of abnormal systemic or intracranial hemorrhage; History of coagulation dysfunction: PLT < 100,000/μl, PT > 14 sec or PTT > 36 sec, and INR > 1.3; Use of anticoagulants (such as warfarin) or antiplatelet drugs (such as aspirin) within one week before surgery, or use of drugs that can increase the risk of bleeding (such as bevacizumab) within one month before focused ultrasound surgery; The subject has cerebrovascular diseases, including but not limited to: intracranial aneurysm, dural arteriovenous malformation (AVM), stroke, intracranial atherosclerotic disease, dural arteriovenous fistula (AVF), etc.; The subject has a brain tumor; The subject has severe abnormal brain structure; Previous corpus callosotomy, VNS, DBS, or stereotactic ablation; Implants in the skull or intracranial cavity; More than 30% of the head area through which the ultrasound irradiation path passes is covered by scars/scalp diseases (such as eczema) or scalp atrophy; The subject has a history of claustrophobia; The overall Skull Density Ratio (SDR) calculated by the subject during screening is less than 0.40 (±0.05); Unable to tolerate the long-term supine and stationary posture required during treatment (about 2-3 hours); Currently participating in another clinical research project; Unable to communicate with researchers and treatment staff; The subject is considered unsuitable for surgery or the study, which may include but is not limited to the following situations: the researcher deems that the subject has any medical, social, or psychological problems that may complicate the evaluation of the study process; The subject had suicidal thoughts within one month before enrollment; The subject has a clinically significant neurological disease other than epilepsy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety | From enrollment to the end of treatment at 1 year
  Evaluate the incidence of adverse events (AEs) within 2 years after treatment with the investigational medical device.

SECONDARY OUTCOMES:
Efficacy | From enrollment to the end of treatment at 1 year
  The efficacy evaluation indicator is the frequency of epileptic seizures, and the data are collected through the epilepsy seizure diary. Quality of life will be measured using the Quality of Life in Epilepsy Inventory-31 (QOLIE-31).

IPD SHARING:
Plan to Share IPD: No